CLINICAL TRIAL: NCT00325598
Title: Partial Breast Irradiation (PBI) for Selected Patients With Early Breast Cancer: A Phase I/II Feasibility Study
Brief Title: Partial Breast Irradiation (PBI) for Selected Patients With Early Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-1053 / 201103235
Record Dates: First submitted 2006-05-12; First posted 2006-05-15 (Estimated); Results first posted 2016-11-07 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Cohort 1 (36 Gy) (Experimental): 36 Gy in 9 fractions BID x 4 1/2 treatment days
  Interventions: Radiation: Partial Breast Irradiation (PBI)
- Cohort 2 (40 Gy) (Experimental): 40 Gy in 10 fractions BID over 5 treatment days
  Interventions: Radiation: Partial Breast Irradiation (PBI)

INTERVENTIONS:
Radiation: Partial Breast Irradiation (PBI)

SUMMARY:
This study investigates the feasibility and safety of delivering radiation therapy only to part of the breast, (the tumor bed and selected areas) rather than the whole breast, for patients with early stage breast cancer.

ELIGIBILITY:
Inclusion Criteria

1. Histologic Documentation:

   * Patients will have histologically confirmed Unicentric Stage I (T1 N0 M0) invasive ductal breast cancer.
   * Histologically negative tumor margin 2 mm or more from any inked edges, or no tumor in a re-excision specimen or final shaved specimen.
   * Tubular, mucinous and medullary variant histologies of infiltrating ductal carcinoma are permitted.
   * Low-grade DCIS (I and II) of 2 cm or less with histologically negative margins of at least 2 mm margins (or a negative re-excision) are permitted.
   * Women age 70 years or older with T1 invasive ductal carcinoma which are estrogen-receptor positive (ER+) with clinically negative axillary nodes who do not undergo surgical lymph node evaluation are also eligible if patient will take hormonal therapy.
   * Patients with T1N0 (i+) tumors on sentinel lymph node mapping or dissection (i.e. is tumor deposit is 0.2mm or less, regardless of whether the deposit is detected by IHC or H&E staining) will also be eligible, provided that completion axillary dissection has been performed to confirm N0 status.
   * In the case where invasive cancer is present, the invasive cancer's pathology will be used regardless if DCIS is also present.
2. Prior Treatment: Patient may have been treated with adjuvant chemotherapy. Patients may be on adjuvant hormonal therapy or begin hormonal therapy following XRT at the discretion of the medical oncologist.

   Radiation therapy should begin within:
   * 4-12 weeks from definitive surgical procedure
   * 2-6 weeks after chemotherapy, if chemotherapy given first
   * Radiation cannot be delivered concurrently with chemotherapy.
3. Age >= 18 years of age
4. ECOG Performance Status 0-2.
5. Signed Informed Consent

Exclusion Criteria

The following guidelines are to assist physicians in selecting patients for whom protocol therapy is safe and appropriate. Physicians should recognize that the following may seriously increase the risk to the patient entering this protocol. Patients who meet the following criteria should not be entered in this study:

1a Multicentric IDC of the breast defined as discontiguous tumors separated by at least 5 cm of uninvolved tissue; alternatively, discontiguous tumors that are clinically or mammographically within separate breast quadrants or subareolar central region.

1. b Multifocal IDC of the breast, defined as discontiguous discrete foci of invasive carcinoma, separated by uninvolved intervening tissue, but within an overall span of 5cm, or within the same breast quadrant or subareolar central region.
2. Tumor > 2.0 cm, nodal involvement on H&E staining, or metastatic involvement
3. Histological evidence of:

   1. Lymphovascular invasion: as defined by a tumor embolus present in an endothelial-lined space; cases with tumor emboli present in a space not lined by endothelial cells but otherwise very suspicious for an angiolymphatic space were also considered ineligible.
   2. EIC (Extensive Intraductal Component): defined as the presence of intraductal carcinoma both within the primary infiltrating ductal tumor (comprising at least 25% of the tumor area) and intraductal carcinoma present clearly beyond the edges of the invasive tumor, or as a predominantly intraductal tumor with one or more areas of focal invasion 7, 55.
   3. Invasive Lobular Carcinoma
   4. Infiltrating carcinoma with mixed ductal and lobular features: cases with ambiguous or mixed histologic features that showed positive E-cadherin staining throughout the tumor by immunohistochemistry were classified as ductal type and considered eligible 56, 57.
   5. Infiltrating papillary carcinoma
   6. Margins: In-situ or invasive carcinoma present less than 2 mm from the inked resection margin.
4. History of cosmetic or reconstructive breast surgery
5. Psychiatric illness which would prevent the patient from giving informed consent. Medical condition such as uncontrolled infection (including HIV), uncontrolled diabetes mellitus or connective tissue diseases (lupus, systemic sclerosis or other collagen vascular diseases) which, in the opinion of the treating physician, would make this protocol unreasonably hazardous for the patient.
6. Patients with a "currently active" second malignancy other than non-melanoma skin cancers. Patients are not considered to have a "currently active" malignancy if they have completed therapy and considered by their physician to be at less than 5% risk of relapse within three years.
7. Patients with diffuse (> 1 quadrant or > 5cm) suspicious microcalcifications
8. Women who are pregnant.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-02-14 (Actual); Primary Completion 2013-04-16 (Actual); Study Completion 2017-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Imran Zoberi, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to participant enrollment on 02/14/2006 and closed to participant enrollment on 04/11/2012.
Groups:
- Cohort 1 (36 Gy): 36 Gy in 9 fractions BID x 4 1/2 treatment days
  Partial Breast Irradiation (PBI)
- Cohort 2 (40 Gy): 40 Gy in 10 fractions BID over 5 treatment days
  Partial Breast Irradiation (PBI)
Period: Overall Study
Arm/Group | Cohort 1 (36 Gy) | Cohort 2 (40 Gy)
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (36 Gy) | Cohort 2 (40 Gy) | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Median (Full Range); unit: years] | 56.5 [36 to 83] | 59 [46 to 76] | 58 [36 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 50 | 100
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of PBI Directed External Radiotherapy as Measured by Percentage of Participants Achieving a Dosimetrically Satisfactory Treatment Plan
Description: -The study will be deemed infeasible if more than 4 patients cannot be given treatment because her tumor is such that a dosimetrically satisfactory treatment plan cannot be devised for her.
Time Frame: Within 1 year of protocol registration
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 (36 Gy) | Cohort 2 (40 Gy)
Number analyzed (Participants) | 50 | 50
percentage of participants | 100 | 100

2. Primary Outcome: Feasibility of PBI Directed External Radiotherapy as Measured by Development of Histological Fat Necrosis or Other Grade 4 Skin or Grade 4 Subcutaneous Toxicity, or Requires Surgery for the Skin/Subcutaneous Toxicity
Description: -The study will be deemed infeasible if more than 4 patients develop histological fat necrosis or other grade 4 skin or grade 4 subcutaneous toxicity, or requires surgery for her skin or subcutaneous toxicity
Time Frame: Within 1 year of protocol registration
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 (36 Gy) | Cohort 2 (40 Gy)
Number analyzed (Participants) | 50 | 50
percentage of participants | 0 | 4

3. Secondary Outcome: Incidence and Severity of Cutaneous Toxicity
Description: * Uses RTOG/EORTC Late Radiation Morbidity Scoring Scheme
  * Grade 0 = none
  * Grade 1 = slight atrophy; pigmentation change; some hair loss
  * Grade 2 = patch atrophy; moderate telangiectasia; total hair loss
  * Grade 3 = marked atrophy; gross telangiectasia
  * Grade 4 = ulceration
  * Worst cutaneous toxicity grade is noted
Time Frame: Up to 5 years
Population: 2 patients in Cohort 1 were not evaluable for this outcome measure because 1 patient withdrew consent and 1 patient was lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (36 Gy) | Cohort 2 (40 Gy)
Number analyzed (Participants) | 48 | 50
Participants
  Grade 0 | 4 | 0
  Grade 1 | 30 | 22
  Grade 2 | 12 | 19
  Grade 3 | 2 | 9
  Grade 4 | 0 | 0

4. Secondary Outcome: Incidence of Breast Fibrosis
Time Frame: Up to 5 years
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (36 Gy) | Cohort 2 (40 Gy)
Number analyzed (Participants) | 48 | 50
Participants | 36 | 39

5. Secondary Outcome: Incidence of Fat Necrosis
Description: -Fat necrosis typically causes a painless mass located superficially in the breast, accompanied by retraction or dimpling of the overlying skin. The skin may be thickened clinically and radiologically. Fat necrosis is firm and relatively circumscribed on palpation. Mammography usually reveals a spiculated, often poorly defined mass that may contain punctate or large, irregular calcifications. Attachment to the skin, dimpling, and thickening of the skin are often evident. Less frequently, the lesion consists of a circumscribed, oil-filled, partly calcified cyst. Early in its development, fat necrosis has the appearance of hemorrhage in indurated fat. After several weeks, the affected area becomes demarcated, forming a distinct yellow-gray and focally reddish tumor. Cystic degeneration may develop in the center of such a lesion, resulting in a cavity that contains oily fluid or necrotic fat.
Time Frame: Up to 5 years
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (36 Gy) | Cohort 2 (40 Gy)
Number analyzed (Participants) | 48 | 50
Participants | 15 | 19

6. Secondary Outcome: Cosmetic Outcome
Description: * Excellent: little or no observable change
  * Good: minimal but identifiable changes
  * Fair: significant results of radiotherapy noted
  * Poor: severe normal tissue sequelae
Time Frame: Up to 5 years
Population: 4 patients in Cohort 1 were not evaluable for this outcome measure because 2 patients did not have the cosmetic outcome performed, 1 patient withdrew consent, and 1 patient was lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (36 Gy) | Cohort 2 (40 Gy)
Number analyzed (Participants) | 46 | 50
Participants
  Excellent | 6 | 11
  Good | 30 | 32
  Fair | 9 | 3
  Poor | 1 | 4

7. Secondary Outcome: Local Control Rate
Description: -Local control rate for this study is the number of participants who remained free of disease in their breast.
Time Frame: Up to 5 years
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (36 Gy) | Cohort 2 (40 Gy)
Number analyzed (Participants) | 48 | 50
Participants | 48 | 50

8. Secondary Outcome: Regional Control Rate
Description: -Regional control rate for this study is the number of participants who remained free from disease in the regional lymph nodes. The regional lymph nodes are the axilla, infraclavicular, supraclavicular, and internal mammary lymph node beds
Time Frame: Up to 5 years
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (36 Gy) | Cohort 2 (40 Gy)
Number analyzed (Participants) | 48 | 50
Participants | 48 | 50

9. Secondary Outcome: Distant Control Rate
Description: -Distant control rate for this study is the number of participants who remained free of cancer at distant sites which is defined as all parts of the body that are not the ipsilateral breast or ipsilateral regional lymph nodes.
Time Frame: Up to 5 years
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (36 Gy) | Cohort 2 (40 Gy)
Number analyzed (Participants) | 48 | 50
Participants | 48 | 50

ADVERSE EVENTS:
Groups:
- Cohort 1 (36 Gy) Acute Toxicities; Cohort 1 (36 Gy) Late Toxicities: 36 Gy in 9 fractions BID x 4 1/2 treatment days
  Partial Breast Irradiation (PBI)
  Follow toxicities from Day 1 through Day 90
- Cohort 2 (40 Gy) Acute Toxicities; Cohort 2 (40 Gy) Late Toxicities: 40 Gy in 10 fractions BID over 5 treatment days
  Partial Breast Irradiation (PBI)
  Follow toxicities from Day 91 through end of follow-up
Arm/Group | Cohort 1 (36 Gy) Acute Toxicities | Cohort 1 (36 Gy) Late Toxicities | Cohort 2 (40 Gy) Acute Toxicities | Cohort 2 (40 Gy) Late Toxicities
Serious Adverse Events (participants affected / at risk) | 3/50 | 0/50 | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 21/50 | 50/50 | 50/50 | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (36 Gy) Acute Toxicities (N=50) | Cohort 1 (36 Gy) Late Toxicities (N=50) | Cohort 2 (40 Gy) Acute Toxicities (N=50) | Cohort 2 (40 Gy) Late Toxicities (N=50)
Breast pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Infection (mastitis) (Infections and infestations) | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Breast edema (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Fever (General disorders) | 1 | 0 | 0 | 0
Rigors/chills (General disorders) | 1 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Costochondritis (General disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (36 Gy) Acute Toxicities (N=50) | Cohort 1 (36 Gy) Late Toxicities (N=50) | Cohort 2 (40 Gy) Acute Toxicities (N=50) | Cohort 2 (40 Gy) Late Toxicities (N=50)
ALT (Investigations) | 0 | 2 | 1 | 3
AST (Investigations) | 0 | 3 | 0 | 1
Abdominal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Agitation (Psychiatric disorders) | 0 | 0 | 4 | 2
Alkaline phosphatase (Investigations) | 0 | 1 | 0 | 1
Allergic reaction/hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 1 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0
Back/sacral pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Blurred vision (Eye disorders) | 0 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Breast assymmetry (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Breast function/lactation (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Breast pain (Reproductive system and breast disorders) | 2 | 14 | 25 | 25
Breast volume/hypoplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Bruising (in absence of Grade 3/4 thrombocytopenia) (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Cardiac conduction abnormality NOS (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac ischemia/infarction (Cardiac disorders) | 0 | 2 | 0 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 5
Chest/shoulder pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0
Cholesterol, serum-high (Investigations) | 0 | 3 | 1 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Creatinine (Investigations) | 0 | 3 | 0 | 1
Depression (Psychiatric disorders) | 0 | 3 | 2 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Dry eye syndrome (Eye disorders) | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dyspareunia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 2 | 2
Edema - Nipple/Areolar (General disorders) | 1 | 2 | 1 | 1
Edema - breast (General disorders) | 2 | 5 | 10 | 10
Edema: arm (General disorders) | 0 | 1 | 0 | 0
Edema: extremity (General disorders) | 0 | 0 | 0 | 1
Edema: limb (General disorders) | 0 | 1 | 2 | 5
Edema: trunk (General disorders) | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 3 | 3 | 15 | 2
Extremity pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Fatigue (General disorders) | 2 | 6 | 12 | 5
Fibrosis - cosmesis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 11 | 8
Fibrosis - deep connective tissue (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Fibrosis/induration (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 2
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hair loss/alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 3
Headache (Nervous system disorders) | 0 | 1 | 0 | 1
Heartburn/dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Hemoglobin (Blood and lymphatic system disorders) | 0 | 2 | 3 | 2
Hemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hot flashes/flushes (Vascular disorders) | 0 | 5 | 8 | 9
Hyperbilirubinemia (Investigations) | 0 | 0 | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 3 | 2 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 4
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 3 | 3 | 26 | 17
Hypertension (Vascular disorders) | 0 | 0 | 1 | 4
Hypertriglyceridemia (Investigations) | 0 | 2 | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypokalemia (Investigations) | 0 | 0 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 3
Hyponatremia (Investigations) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Infection with unknown ANC - bronchus (Infections and infestations) | 0 | 1 | 0 | 0
Infection with unknown ANC - ungual (Infections and infestations) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 4 | 3
Joint function (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2
Joint pain (Musculoskeletal and connective tissue disorders) | 0 | 5 | 3 | 9
Left ventricular diastolic dysfunction (Cardiac disorders) | 0 | 1 | 0 | 0
Leukocytes (Investigations) | 0 | 0 | 1 | 2
Libido (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Limb pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Lymphopenia (Investigations) | 0 | 1 | 5 | 6
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 3
Muscle pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal - stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Neuropathy: balance (Nervous system disorders) | 0 | 0 | 1 | 1
Neuropathy: cranial - CN VIII hearing and balance (Nervous system disorders) | 0 | 2 | 0 | 0
Neuropathy: cranial - CN VIII sensory-taste (Nervous system disorders) | 0 | 0 | 1 | 0
Neuropathy: motor (Nervous system disorders) | 0 | 0 | 1 | 0
Orgasmic dysfunction (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 1
Platelets (Investigations) | 0 | 1 | 0 | 1
Pneumonitis (Infections and infestations) | 0 | 0 | 0 | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 2
Rash: dermatitis associated with radiation (Injury, poisoning and procedural complications) | 0 | 1 | 21 | 3
Rib tenderness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Rigors/chills (General disorders) | 0 | 0 | 0 | 2
Sensory neuropathy (Nervous system disorders) | 0 | 0 | 2 | 1
Seroma (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Sweating (diaphoresis) (General disorders) | 0 | 3 | 4 | 1
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 1
Throat pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Thrombosis/thrombus/embolism (Vascular disorders) | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1
Unknown skin - Skin (cellulitis) (Infections and infestations) | 0 | 0 | 1 | 1
Urinary frequency/urgency (Renal and urinary disorders) | 0 | 1 | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 1 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Vaginal dryness (Reproductive system and breast disorders) | 0 | 2 | 0 | 2
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Vaginal pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Valvular heart disease (Cardiac disorders) | 0 | 1 | 0 | 0
Voice changes (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Watery eye (Eye disorders) | 0 | 0 | 0 | 1
Wound complication, non-infectious (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes